CLINICAL TRIAL: NCT01833286
Title: Radiofrequency Ablation Combined With Transcatheter Arterial Chemoembolization Versus Re-resection for Recurrent Hepatocellular Carcinoma
Brief Title: TACE+RFA Versus Re-resection for Recurrent Small Hepatocellular Carcinoma
Acronym: TACE-RFA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACE+RFA VS. Re-resection; 5010 (Other: the 5010 Foundation of Sun Yat-sen University)
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma; Surgery; Ablation
Keywords: hepatocellular carcinoma; repeat hepatectomy; radiofrequency ablation; transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE+RFA (Experimental): TACE was performed according to the following protocol: All patients underwent a distal super-selective catheterization of the hepatic arteries using a coaxial technique and micro-catheters (2.9 Fr, Terumo Corporation, Tokyo, Japan). Then, the same three chemotherapeutic agents at the same dosages were used throughout this study, regardless of tumor number and size. Hepatic artery infusion chemotherapy was performed using carboplatin 300 mg. After that, chemolipiodolization was performed using epirubicin 50 mg, and mitomycin C 8 mg mixed with 5 mL of lipiodol. If the territory of the chemolipiodolized artery did not show stagnant flow, pure lipiodol was then injected. RFA was performed after TACE in 2 months by using a commercially available system (RF 2000; Radio-Therapeutics Mountain View, CA), and a needle electrode with a 15 Ga insulated cannula with 10 hook-shaped expandable electrode tines with a diameter of 3.5 cm at expansion (LeVeen; RadioTherapeutics).
  Interventions: Procedure: TACE+RFA
- re-resection (Active Comparator): Re-resection was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant and the possibility of a negative resection margin. We performed anatomical resection aiming at a resection margin of at least 1 cm. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 minutes and 5 minutes, respectively. Hemostasis of the raw liver surface was done with suturing and application of fibrin glue.
  Interventions: Procedure: re-resection

INTERVENTIONS:
Procedure: TACE+RFA — TACE first, followed by RFA within 2 months
  Arms: TACE+RFA
Procedure: re-resection — repeat hepatectomy for recurrent small HCC
  Other Names: repeat hepatectomy
  Arms: re-resection

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Partial hepatectomy is still considered as the conventional therapy for HCC. Intrahepatic recurrence of HCC after partial hepatectomy is common and was reported to be more than 77% within 5 years after surgery. Repeat hepatectomy is an effective treatment for intrahepatic HCC recurrence, with a 5-year survival rate of 19.4-56%. This is comparable to the survival after initial hepatectomy for HCC. Unfortunately, repeat hepatectomy could be carried out only in a small proportion of patients with HCC recurrence (10.4-31%), either because of the poor functional liver reserve or because of widespread intrahepatic recurrence. In the past two decades, percutaneous radiofrequency ablation (PRFA) has emerged as a new treatment modality and has attracted great interest because of its effectiveness and safety for small HCC (≤ 5.0 cm). Studies using PRFA to treat recurrent HCC after partial hepatectomy reported a 3-year survival rate of 62-68%, which is comparable to those achieved by surgery. PRFA is particularly suitable to treat recurrent HCC after partial hepatectomy because these tumors are usually detected when they are small and PRFA causes the least deterioration of liver function in the patients. Our previous retrospective study demonstrated that RFA was comparable to re-resection for recurrent HCC, and our recent RCT showed that RFA combined with TACE is superior to RFA for HCC ≤7.0cm. So our hypothesis is that RFA combined with TACE is superior to re-resection for recurrent small HCC. The aim of this retrospective study is to compare the outcome of reresection with TACE+RFA for small recurrent HCC after partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 75 years;
2. recurrence of HCC 12 months after initial hepatectomy;
3. no other treatment received except for the initial hepatectomy;
4. Single tumor≤5cm in diameter; or 2-3 lesions each ≤ 3.0 cm
5. lesions visible on ultrasound and with an acceptable and safe path between the lesion and the skin as shown on ultrasound;
6. no severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
7. Eastern Co-operative Oncology Group performance(ECOG) status 0 -1

Exclusion Criteria:

1. the presence of vascular invasion or extrahepatic spread on imaging;
2. a Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3), esophageal or gastric variceal bleeding or hepatic encephalopathy;
3. an American Society of Anesthesiologists (ASA) score ≥ 3 -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
disease-free survival | 5 year

OTHER OUTCOMES:
Mortality | 30 days
Morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: minshan chen, M.D., Principal Investigator — Department of Hepatobiliary Surgery, Sun Yat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991
- [Background] Peng ZW, Zhang YJ, Liang HH, Lin XJ, Guo RP, Chen MS. Recurrent hepatocellular carcinoma treated with sequential transcatheter arterial chemoembolization and RF ablation versus RF ablation alone: a prospective randomized trial. Radiology. 2012 Feb;262(2):689-700. doi: 10.1148/radiol.11110637. Epub 2011 Dec 12. PMID 22157201
- [Background] Peng ZW, Guo RP, Zhang YJ, Lin XJ, Chen MS, Lau WY. Hepatic resection versus transcatheter arterial chemoembolization for the treatment of hepatocellular carcinoma with portal vein tumor thrombus. Cancer. 2012 Oct 1;118(19):4725-36. doi: 10.1002/cncr.26561. Epub 2012 Feb 22. PMID 22359112
- [Derived] Zhang YJ, Chen J, Zhou Z, Hu D, Wang J, Pan Y, Fu Y, Hu Z, Xu L, Chen MS. Transarterial Chemoembolization with Radiofrequency Ablation versus Surgical Resection for Small Late-Recurrence Hepatocellular Carcinoma. Radiology. 2025 Feb;314(2):e241096. doi: 10.1148/radiol.241096. PMID 39903071